CLINICAL TRIAL: NCT02805894
Title: A Phase I-II Dose-escalation Study of NBTXR3 Activated by EBRT or EBRT With Brachytherapy in Patients With Newly Diagnosed Unfavorable Intermediate or High Risk Prostate Adenocarcinoma Treated With Androgen Deprivation
Brief Title: NBTXR3 Nanoparticles and EBRT or EBRT With Brachytherapy in the Treatment of Prostate Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Prostate cancer treatment has greatly changed since the initiation of this trial and therefore we have stopped this trial to allow for further evaluation of the treatment landscape
Sponsor: Nanobiotix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBTXR3-104
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NBTXR3 activated by IMRT only (Experimental): Part I Dose Escalation
  NBTXR3 will be administered by intra-prostate injection and then activated 10 days later by:
  - EBRT delivered as 45 Gy in 25 fractions of 1.8 Gy each; to the prostate and seminal vesicles, followed by 34.2 Gy in 19 fractions to the prostate and proximal seminal vesicles , over 9-10 weeks, utilizing intensity modulated radiotherapy (IMRT) with daily image guidance aligned to implanted fiducial markers (COHORT A)
  Interventions: Drug: NBTXR3 activated by IMRT only
- NBTXR3 activated by Brachytherapy & IMRT (Experimental): Part I Dose Escalation
  NBTXR3 will be administered by intra-prostate injection and then activated 10 days later by:
  - Brachytherapy Boost and EBRT delivered as a single fraction of 15 Gy in one day to the prostate by High Dose Rate Brachytherapy followed by EBRT (initiated within 2-4 weeks after completion of Brachytherapy), delivered as 45 Gy in 25 fractions of 1.8 Gy to the prostate and seminal vesicles utilizing intensity modulated radiotherapy (IMRT) with daily image guidance aligned to implanted fiducial markers (COHORT B)
  Interventions: Drug: NBTXR3 activated by Brachytherapy & IMRT

INTERVENTIONS:
Drug: NBTXR3 activated by IMRT only — Single local administration of NBTXR3 by injection into the prostate gland prior to the IMRT treatment
  Other Names: Hafnium Oxide nanoparticles
  Arms: NBTXR3 activated by IMRT only
Drug: NBTXR3 activated by Brachytherapy & IMRT — Single local administration of NBTXR3 by injection into the prostate gland prior to the Brachytherapy & IMRT treatment
  Other Names: Hafnium Oxide nanoparticles
  Arms: NBTXR3 activated by Brachytherapy & IMRT

SUMMARY:
This study is a Phase 1/2 open-label involving 2 groups of patients newly diagnosed with either unfavorable intermediate risk or high risk prostate adenocarcinoma. One group will receive only EBRT and the other group will receive a Brachytherapy boost and EBRT. Both groups will receive treatment with androgen deprivation. There will be 2 consecutive steps, a dose escalation and a subsequent dose expansion part.

DETAILED DESCRIPTION:
This is a Phase 1/2 prospective, open-label, two cohorts, non-randomized trial consisting of two consecutive steps, a dose escalation and a subsequent dose expansion part.

PART 1 DOSE ESCALATION: subjects with newly diagnosed Unfavorable Intermediate

Risk (UIR) or High Risk (HR) prostate adenocarcinoma, will participate in a dose escalation of NBTXR3 activated by two different radiation schedules. NBTXR3 will be administered by intra-prostate injection and then activated 10 days later either by:

* EBRT delivered as 45 Gy in 25 fractions of 1.8 Gy each; to the prostate and seminal vesicles, followed by 34.2 Gy in 19 fractions to the prostate and proximal seminal vesicles, over 9-10 weeks, utilizing intensity modulated radiotherapy (IMRT) with daily image guidance aligned to implanted fiducial markers (COHORT A) or,
* Brachytherapy Boost and EBRT delivered as a single fraction of 15 Gy in one day to the prostate by High Dose Rate Brachytherapy followed by EBRT (initiated within 2-4 weeks after completion of Brachytherapy), delivered as 45 Gy in 25 fractions of 1.8 Gy to the prostate and seminal vesicles utilizing intensity modulated radiotherapy (IMRT) with daily image guidance aligned to implanted fiducial markers (COHORT B)

PART 2 DOSE EXPANSION: Two parallel cohorts of subjects, A and B, 20 subjects per cohort, will be treated at either the RD1 (Recommended Dose of NBTXR3 given as intraprostate injection and activated by EBRT) or RD2 (Recommended Dose of NBTXR3 given as intra-prostate injection and activated by Brachytherapy Boost and EBRT), as determined in the Phase I dose escalation of the trial.

All subjects will receive androgen deprivation therapy (ADT) LHRH / GnRH agonist beginning 8 weeks before the NBTXR3 administration and for 24 months in subjects with (HR) prostate adenocarcinoma. The duration of ADT in subjects with (UIR) disease will be of 6 months.

Subjects will receive a single intra-prostate injection of NBTXR3 which will be delivered to the prostate via transperineal injection under TRUS guidance injection. NBTXR3 injection will be performed on Day 1 and will be assessed for safety, intra-prostate availability and presence of NBTXR3 in the peripheral circulation.

COHORT A: External beam radiation therapy will be delivered to the prostate starting within 9 days after the NBTXR3 injection (Day 10). Total dose of 79.2 Gy, delivered as 25 fractions of 1.8 Gy to the prostate and seminal vesicles (45 Gy), followed by 34.2 Gy in 19 fractions to the prostate and proximal seminal vesicles, delivered over 9-10 weeks, utilizing intensity modulated radiotherapy (IMRT) with daily image guidance aligned to implanted fiducial markers COHORT B: HDR Brachytherapy implantation will be performed within 9 days after NBTXR3 injection (Day 10). Brachytherapy Boost delivered as a single fraction of 15 Gy in one day to the prostate by High Dose Rate Brachytherapy followed by EBRT (initiated within 2-4 weeks after completion of Brachytherapy) delivered as 45 Gy in 25 fractions of 1.8 Gy to the prostate and seminal vesicles utilizing intensity modulated radiotherapy (IMRT) with daily image guidance aligned to implanted fiducial markers.

Subjects will be followed for safety assessment until the end of the study. Before the onset of study treatment, subjects must have a histologic diagnosis of either Unfavorable Intermediate Risk (UIR) or High Risk (HR) prostate adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Histologically confirmed adenocarcinoma of the prostate gland by needle core samples with assigned Gleason score
* Subjects ADT naive or subjects who are already on ADT treatment and scheduled to receive radiation therapy for their adenocarcinoma of prostate are eligible. An 8-week course of ADT is required to be completed prior to NBTXR3 administration and initiation of radiation therapy.
* Pelvic and para-aortic lymph nodes must be negative on CT-scan or MRI of the abdomen and pelvis performed within 12 weeks prior to enrollment into the study
* Prostate adenocarcinoma with High Risk (HR) and Unfavorable Intermediate Risk (UIR) for recurrence classification as determined by one of the following combinations:

  * High risk (HR): subjects with one or more of the following risk factors:

    * Clinical stage: T3/T4
    * Gleason score (GS): 8-10
    * PSA > 20
    * N0
  * Unfavorable Intermediate Risk (UIR): subjects with no HR features but with one or more of the following adverse risk factors:

    * At least 2 of the following 3 factors: Gleason score(GS) 3+4=7 and/or PSA 10-20 and/or T2b/c
    * Gleason score (GS) 4+3=7
    * Greater than 50% of biopsy cores positive and at least one other risk factor:

Gleason score (GS) 7 and/or PSA 10-20 and/or T2b/c

* No evidence of bone metastases (M0) on bone scan within 120 days prior to registration (PET/CT is an acceptable substitute). Equivocal bone scan findings are allowed if bone CT or MRI of hot spots are negative for metastasis
* Baseline serum PSA value performed with an FDA-approved assay within 120 days prior to registration. Study entry PSA should not be obtained within 10-day period following prostate biopsy or following initiation of hormonal therapy
* ECOG performance status must be 0 or 1
* Adequate function of bone marrow:

  * Hemoglobin > 100 g/L
  * Absolute Neutrophils > 1.5 x 109/L
  * Platelets > 100 x 109/L,
* Adequate function of kidney:

  * Serum creatinine < 1.5 x ULN
* Adequate function of liver:

  * AST ≤ 3.0 x ULN
  * ALT ≤ 3.0 x ULN
  * Total bilirubin ≤ 1.5 x ULN
* Non-Childbearing Potential: Male subjects and their partners must meet one of the following criteria to be considered of non-childbearing potential:

  * Males have undergone sterilization with appropriately confirmed absence of sperm in the post-vasectomy ejaculate, or
  * Heterosexually active males and their partners of childbearing potential must agree or use at least 2 forms of highly effective methods of contraception, including at least 1 barrier method. Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of <1% per year when used consistently and correctly (i.e., perfect use). Contraception must include male condom or female condom used with a spermicide (i.e., foam, gel, film, cream, suppository) as well as established use of oral, injected or implanted hormonal methods of contraception, correctly placed intrauterine device or intrauterine system.

Exclusion Criteria:

* Written Informed Consent not obtained, signed and dated
* History of colorectal surgery, or repeated endoscopic examinations/interventions related to anorectal diseases or proximal urethral stricture requiring dilatation
* Prostate size volume ≥90 cc
* Brachytherapy with EBRT in subjects whose prostate volume is >60cc
* Severe, active co-morbidity, defined as follows:

  * Inflammatory bowel disease, active rectal diverticulitis, Crohn's disease affecting the rectum, anal stenosis or ulcerative colitis. (Nonactive diverticulitis and Crohn's disease not affecting the rectum are allowed)
  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of randomization
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC (Centers for Disease Control) definition
* Prior invasive malignancy, except non-melanoma skin cancer, carcinoma in-situ of the bladder or head and neck region, unless disease free for a minimum of 2 years
* Subjects with congenital long QT syndrome or subjects taking Class IA, Class III or Class IC anti-arrhythmic medications will require a cardiologist's evaluation prior to eligibility assessment. subjects with cardiovascular diseases can be included as long as the benefits of androgen deprivation therapy outweigh the potential risk of cardiovascular events
* Uncontrolled lung disease
* Subjects with any evidence of distant metastases
* subjects with any contraindication to pelvic radiotherapy including, but not limited to, previous pelvic radiotherapy or brachytherapy
* Presence of bilateral hip replacement prostheses
* Hormonal therapy (luteinizing hormone-releasing hormone [LHRH] agonist or oral anti-androgen) exceeding 4 months prior to registration
* Declared high-risk for anesthesia by attending anesthesiologist, cardiologist, or other physician
* Complete initial work up earlier than 12 weeks prior to subject registration
* Subjects unable to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Subjects participating in another clinical investigation at the time of signature of the informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and early Dose Limiting Toxicities (DLT) of NBTXR3 | 24 months
Recommended Dose(s) of NBTXR3 | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dicker, MD, Principal Investigator — Thomas Jefferson University Hospital Philadelphia, PA
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute/Brigham and Women's Hospital, Boston, Massachusetts
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No